CLINICAL TRIAL: NCT03395847
Title: A Pilot Study of Pembrolizumab Monotherapy in Patients With Previously Treated Advanced Gastroesophageal Adenocarcinoma
Brief Title: Pembrolizumab in Treating Patients With Metastatic or Unresectable Gastroesophageal Adenocarcinoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0905; NCI-2018-00946 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0905 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-11-30; First posted 2018-01-10 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Advanced Gastroesophageal Junction Adenocarcinoma; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Gastric Cancer AJCC v8; Clinical Stage IVB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVB Gastric Cancer AJCC v8; Gastroesophageal Junction Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Pathologic Stage IV Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IV Gastric Cancer AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Gastric Cancer AJCC v8; Postneoadjuvant Therapy Stage IV Gastric Cancer AJCC v8; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This early phase I trial studies how well pembrolizumab works in treating patients with gastroesophageal adenocarcinoma that has spread to other places or cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall response rate (ORR) of intravenous administration of pembrolizumab by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in adult subjects with advanced (unresectable and/or metastatic) and previously treated gastroesophageal adenocarcinoma.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response (DOR), disease control rate (DCR), time to progression (TTP), progression-free survival (PFS), and overall survival (OS) using RECIST 1.1 and immune-related (ir)RECIST criteria.

II. To perform exploratory biomarkers to study the correlation between immunological and molecular changes in tumor tissues and peripheral blood with clinical outcomes (DOR, DCR, TTP, PFS, and OS) using RECIST 1.1, and irRECIST rate of adverse events.

III. To determine the safety and tolerability of intravenous administration of pembrolizumab or pembrolizumab plus ramucirumab in adult subjects with advanced (unresectable and/or metastatic) and previously treated gastroesophageal adenocarcinoma.

EXPLORATORY OBJECTIVES:

I. To explore the association between PD-L1 expression by immunohistochemistry, shed PD-L1 levels, somatic gene expression profiling and antitumor efficacy of pembrolizumab based on RECIST 1.1 imaging criteria as well as overall survival.

II. To explore the relationship between genomic variation and response to the treatment administered.

III. Tissue and blood immune monitoring will be conducted through our immune platform group as detailed per the biomarker section based on 3 biopsies done at the following time points: 1) pre-treatment, 2) 6 weeks after therapy, and 3) and an optional biopsy upon progression.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The subject (or legally acceptable representative if applicable) provides written informed consent for the trial. The subject may also provide consent for future biomedical research. However the subject may participate in the main trial without participating in future biomedical research.
* Be willing and able to provide written informed consent/assent for the trial.
* Histologically and cytologically documented diagnosis as gastroesophageal adenocarcinoma.
* Have a documented advanced (metastatic and/or unresectable) gastroesophageal adenocarcinoma that is incurable and for which prior first-line or later-line standard of care (SOC) treatments have failed. There is no limit to the number of prior treatment regimens. Prior neoadjuvant or adjuvant therapy included in initial treatment may not be considered first- or later-line SOC treatment unless such treatments were completed less than 12 months prior to the current tumor recurrence.
* Have submitted an evaluable tissue sample for biomarker analysis from a newly obtained endoscopic, core, incisional, or excisional biopsy of a tumor lesion not previously irradiated. The tumor tissue submitted for analysis must be from a single tumor tissue specimen and of sufficient quantity and quality to allow biomarker study. A newly obtained tumor specimen, defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1, for biomarker characterization will be required for enrollment of all subjects. Tissue from tumor progressing at a site of prior radiation may be allowed for biomarker characterization upon agreement from Merck. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Merck.
* Have measurable disease based on RECIST 1.1 as assessed by the investigator. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Life expectancy of greater than 3 months per the judgment of the investigators.
* Absolute neutrophil count (ANC) >= 1,500 /mcL (within 5 days prior to the start of study treatment).
* Platelets >= 100,000/mcL (within 5 days prior to the start of study treatment).
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (within 5 days prior to the start of study treatment).
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional upper limit of normal (ULN) (within 5 days prior to the start of study treatment). Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 5 days prior to the start of study treatment).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (within 5 days prior to the start of study treatment).
* Albumin: >= 2.5 mg/dL (within 5 days prior to the start of study treatment).
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 5 days prior to the start of study treatment).
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 5 days prior to the start of study treatment).
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Male and female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating in or has participated in a study of an investigational agent or used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Subjects who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has severe hypersensitivity (>= grade 3) to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with =< grade 2 neuropathy or alopecia are an exception to this criterion.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention as determined by the investigators prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiological stable (i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to the first dose of trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required treatment with steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (TCR) (e.g., CTLA-4, OX 40, CD137).
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies). No HIV testing is required unless mandated by local health authority.
* Had a solid organ or hematologic transplant.
* Has a known history of hepatitis B virus (HBV; hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV; HCV ribonucleic acid [RNA] [qualitative] is detected) infection. No testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
* Has received a live vaccine within 30 days prior to the first dose of the trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette - Guerin (BCG), and typhoid vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 4 years
  Defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR). Responses are based on assessments by the blinded MD Anderson radiology per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Exact method based on binomial distribution (Clopper-Pearson method).

SECONDARY OUTCOMES:
Duration of response | From first documented evidence of CR or PR up to 4 years
  Based on assessments by MD Anderson radiology per RECIST 1.1. Summary statistics using Kaplan-Meier method, if sample size permits.
Disease control rate | Up to 4 years
  Defined as the percentage of subjects who have achieved CR, PR, or stable disease (SD) for at least 24 weeks based on assessments by MD Anderson radiology per RECIST 1.1. Exact method based on binomial distribution (Clopper-Pearson method).
Time to progression | From the first day of study treatment up to 4 years
  Assessed per RECIST 1.1 based on assessments by MD Anderson radiology. Summary statistics using Kaplan-Meier method.
Progression-free survival per RECIST 1.1 based on assessments by MD Anderson radiology | From the first day of study treatment to the first documented disease progression up to 4 years
  Summary statistics using Kaplan-Meier method.
Overall survival | From first dose of study medication up to 4 years
  Summary statistics using Kaplan-Meier method.
Incidence of adverse events | Up to 30 days post treatment
  Defined by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Adverse events will be assessed. Specific events will be collected and designated as events of clinical interest (ECIs).

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A Ajani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org